CLINICAL TRIAL: NCT03195088
Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Rising Subcutaneous Doses of BI 473494 in Healthy Male Subjects (Single-blind, Partially Randomised, Placebo-controlled Parallel Group Design)
Brief Title: Evaluation of Safety and Tolerability of Single Rising Doses of BI 473494 in Healthy Subjects
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated (Business Reasons)
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1400-0001; 2016-003224-24 (EudraCT Number)
Record Dates: First submitted 2017-06-20; First posted 2017-06-22 (Actual); Results first posted 2022-06-22 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Healthy participants were administered a single dose of placebo matching BI 473494 solution via subcutaneous injection.
  Interventions: Drug: Placebo
- BI 473494 35 μg (Experimental): Healthy participants were administered a single dose of 35 micrograms (μg) BI 473494 solution via subcutaneous injection.
  Interventions: Drug: BI 473494
- BI 473494 75 μg (Experimental): Healthy participants were administered a single dose of 75 micrograms (μg) BI 473494 solution via subcutaneous injection.
  Interventions: Drug: BI 473494

INTERVENTIONS:
Drug: BI 473494 — Solution for injection
  Arms: BI 473494 35 μg; BI 473494 75 μg
Drug: Placebo — Solution for injection
  Arms: Placebo

SUMMARY:
The primary objective of this trial is to investigate the safety and tolerability of single rising doses of BI 473494 in healthy male subjects.

The secondary objective is the exploration of PK including dose proportionality, and PD of BI 473494 after single dosing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, based on a complete medical history including a physical examination, vital signs (Blood Pressure [BP], Pulse Rate [PR]), 12-lead Electrocardiogram [ECG], and clinical laboratory tests
* Age of 18 to 45 years (incl.)
* Body Mass Index [BMI] of 20.0 to 29.9 kg/m2 (incl.)
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice [GCP] and local legislation

Exclusion Criteria:

* Any finding in the medical examination (including Blood Pressure [BP], Pulse Rate [PR] or Electrocardiogram [ECG]) is deviating from normal and judged as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 bpm
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease judged as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Use of drugs within 30 days prior to administration of trial medication if that might reasonably influence the results of the trial (incl. QT/QTc interval prolongation)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* Further exclusion criteria apply

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: It was planned to include healthy participants in this single-rising dose trial with a single-blind, partially randomised, placebo controlled and parallel group design. They were recruited from the volunteer's pool of the study site.
Pre-assignment Details: All participants were screened for eligibility to participate in the trial by the trial site. The site ensured that the participants met all strictly implemented inclusion/exclusion criteria. Participants were not to be assigned to treatment groups if any one of the specific entry criteria were violated.
Groups:
- Placebo Matching BI 473494: Healthy participants were administered a single dose of placebo matching BI 473494 solution via subcutaneous injection.
Period: Overall Study
Arm/Group | Placebo Matching BI 473494 | BI 473494 35 μg | BI 473494 75 μg
Started (Started are treated) | 4 | 6 | 6
Completed | 4 | 6 | 6
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set (TS) : The TS included all subjects who were dispensed study medication and were documented to have taken at least one dose of BI 473494.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Matching BI 473494 | BI 473494 35 μg | BI 473494 75 μg | Total
Number analyzed (Participants) | 4 | 6 | 6 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.3 (5.9) | 34.0 (7.4) | 30.2 (6.8) | 32.6 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 4 | 6 | 6 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 6 | 6 | 16
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 4 | 5 | 6 | 15
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Drug-related Adverse Events (AEs) Analysed as Investigator Defined Drug-related AEs
Description: Percentage of participants with drug-related adverse events (AEs) analysed as investigator defined drug-related AEs is presented. Medical judgment was used to determine the relationship between the AEs and the study medication, considering all relevant factors, including pattern of reaction, temporal relationship, de-challenge or re-challenge, confounding factors such as concomitant medication, concomitant diseases and relevant history.
Time Frame: From drug administration until End of trial (EOT), up to 40 days.
Population: as for baseline characteristics
Measure: Number; unit: Percentage of participants (%)
Arm/Group | Placebo Matching BI 473494 | BI 473494 35 μg | BI 473494 75 μg
Number analyzed (Participants) | 4 | 6 | 6
Percentage of participants (%) | 0.0 | 0.0 | 16.7

2. Secondary Outcome: Area Under the Concentration-time Curve of BI 473494 Over the Time Interval From 0 to the Last Quantifiable Time Point (AUC0-tz)
Description: AUC0-tz, area under the concentration-time curve of BI 473494 over the time interval from 0 to the last quantifiable time point is presented.
Time Frame: Pharmacokinetic samples were taken 1:00 hour:minute (h:m) pre-dose and 3:00, 6:00, 9:00, 12:00, 15:00 , 22:00, 24:00, 28:00, 34:00, 39:00, 48:00, 60:00, 72:00, 96:00, 120:00, 168:00, 240:00, 336:00, 504:00 and 672:00 h:m after drug administration on day 1
Population: Pharmacokinetic (PK) parameter analysis set (PKS): The PKS included all subjects from the TS who received study medication and provided at least one secondary PK parameter that was not excluded due to important protocol deviations with respect to the statistical evaluation of PK endpoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomole*Hours/Litre (nmol*h/L)
Arm/Group | BI 473494 35 μg | BI 473494 75 μg
Number analyzed (Participants) | 6 | 6
Nanomole*Hours/Litre (nmol*h/L) | 162 (24.8) | 546 (18.5)

3. Secondary Outcome: Maximum Measured Concentration of BI 473494 (Cmax)
Description: Cmax, maximum measured concentration of BI 473494 is presented.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanomole/Litre (nmol/L)
Arm/Group | BI 473494 35 μg | BI 473494 75 μg
Number analyzed (Participants) | 6 | 6
Nanomole/Litre (nmol/L) | 0.82 (23.1) | 1.88 (17.5)

ADVERSE EVENTS:
Time Frame: From drug administration until End of trial (EOT), up to 40 days.
Arm/Group | Placebo Matching BI 473494 | BI 473494 35 μg | BI 473494 75 μg
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/6 | 1/6
Other Adverse Events (participants affected / at risk) | 0/4 | 2/6 | 1/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matching BI 473494 (N=4) | BI 473494 35 μg (N=6) | BI 473494 75 μg (N=6)
Acute polyneuropathy (Nervous system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Matching BI 473494 (N=4) | BI 473494 35 μg (N=6) | BI 473494 75 μg (N=6)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 0 | 1
Peripheral coldness (Vascular disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated due to business reasons after the second of 11 planned dose groups. Therefore, only two dose groups were evaluated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2017-05-02): https://cdn.clinicaltrials.gov/large-docs/88/NCT03195088/Prot_002.pdf
  • Statistical Analysis Plan (2019-01-29): https://cdn.clinicaltrials.gov/large-docs/88/NCT03195088/SAP_001.pdf